CLINICAL TRIAL: NCT02667834
Title: Efficiency of the French Translation Program:Social Cognition and Interactive Training (SCIT) of Negative Symptoms in Schizophrenia
Brief Title: Efficiency of the French Translation Social Cognition and Interactive Training (SCIT)Program
Acronym: SCIT-VF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-A00072-45
Record Dates: First submitted 2016-01-19; First posted 2016-01-29 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
Keywords: social cognition; cognitive remediation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Social Cognition and Interaction Training (SCIT) (Experimental): SCIT Social cognition and interaction training program.
  Interventions: Behavioral: Social Cognition and Interaction Training (SCIT)
- Therapeutic education program (ETP) (Active Comparator): Therapeutic education program
  Interventions: Behavioral: therapeutic education program (ETP)

INTERVENTIONS:
Behavioral: Social Cognition and Interaction Training (SCIT) — A randomized, controled trial of social cognition and interaction training ( SCIT) for patients with schizophrenia Spectrum disorders
  Arms: Social Cognition and Interaction Training (SCIT)
Behavioral: therapeutic education program (ETP) — usual treatment ,30 hours with therapist, only discussion between patients
  Arms: Therapeutic education program (ETP)

SUMMARY:
Social cognition and interaction training (SCIT), a group-based treatment that aims to improve both processing social information and functioning, may be an effective treatment for enhancing the social skills of people with schizophrenia. This study will compare the effectiveness of Social cognition and interaction training (SCIT) versus treatment as usual (ETP) in helping people with schizophrenia improve their social cognition and social functioning so specially on negative symptoms. Many studies show a connection between negative symptom and social cognition in schizophrenia.

DETAILED DESCRIPTION:
This is a multicenter (6 centers in France), randomized, controlled trial compared people aged 18 to 50 years with a diagnostic of schizophrenia according to the Diagnostic and Statistical manual of Mental disorders, 4th edition (DSM-IV-TR), the Social Cognition and Interaction Training (SCIT) program will be compared to an already validated neurocognitive remediation program : therapeutic education program (ETP) Social Cognition and Interaction Training (SCIT) is composed of three phases: emotion training, figuring out situations, and integration. Social Cognition and Interaction Training (SCIT) will be delivered by therapists in 20 weekly sessions over 5 months.

160 patients will be randomized as follows: - Arm1, experimental: Social Cognition and Interaction Training (SCIT): 30h with therapist, videos and photos exercises - Arm 2, control: therapeutic education program (ETP): 30h with therapist, only discussion between patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 50 years old
* Diagnosis of schizophrenia according to the DSM-IV-TR
* French speaker
* Unchanged psychotropic treatment during month preceding the inclusion
* Patients having given their consent lit to participate in the study
* Patients not having been part of therapeutic education program during six months preceding the inclusion
* Affiliated to the French social security

Exclusion Criteria:

* Alcohol or drug dependence(according to the DSM-IV-TR),except Tobacco
* History of neurobiological illness or trauma
* Taking of medicine with somatic aim having a cerebral or psychic impact (ex: corticosteroids)
* Simultaneous participation on another program of cognitive remediation
* The ineffectiveness of neuroleptic treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Scale of Assessment of Negative Symptoms | 40 weeks
  Improvement of negative symptoms of schizophrenia in patients who received Social Cognition and Interaction Training (SCIT) program compared to patients receiving a Therapeutic Education Program (ETP), equivalent in number, duration and rhythm of sessions

SECONDARY OUTCOMES:
Change from baseline in positive and negative symptoms scale (PANSS) | 40 weeks
  Scales for clinical and psychosocial functioning measurement

CONTACTS AND LOCATIONS:
Overall Officials: FRANCK NICOLAS, PUPH, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier de Clermont de l'Oise, Clermont, OISE, France

IPD SHARING:
Plan to Share IPD: No